CLINICAL TRIAL: NCT06485635
Title: Real-life-Persistence to Antifibrotic Treatments
Acronym: REPEAT
Status: Active, not recruiting | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0568
Record Dates: First submitted 2024-06-10; First posted 2024-07-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib; pirfenidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a reimbursement of AF treatment
  Interventions: Drug: Nintedanib; Drug: Pirfenidone

INTERVENTIONS:
Drug: Nintedanib — Nintedanib
Drug: Pirfenidone — Pirfenidone

SUMMARY:
This study will help to better understand the persistence rate to antifibrotic (AF) treatment in real life in France and to identify potential areas for improvement by investigating the factors associated with a non-persistence rate to AF treatment.

Primary objective of the study is to measure the percentage of patients still treated up to 30 months after AF treatment initiation.

ELIGIBILITY:
Inclusion criteria:

All patients with a reimbursement of AF treatment between 2018 and 2022 will be included for analysis.

Exclusion criteria:

No exclusion criteria will be applied.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a reimbursement of AF treatment between 2018 and 2022 will be included for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 10646 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Persistence to antifibrotic (AF) treatment (measured as percentage of patients still treated up to 30 months after AF treatment initiation) | up to 30 months

SECONDARY OUTCOMES:
AF prevalence in French population | up to 5 years
AF incidence in French population | up to 4 years
Number of AF treated patients split by indication | up to 2 years
  Indications:
  * Idiopathic Pulmonary Fibrosis (IPF)
  * Interstitial Lung Disease associated with Systemic Sclerosis (SSc-ILD)
  * Progressive Pulmonary Fibrosis (PPF)
Number of patients adherent to AF treatment | up to 30 months
  In incident AF patients, percentage of days covered (PDC) will be calculated at different time point to measure the adherence to AF treatment for patients persistent to treatment at this time point.
  The PDC is the ratio dividing the number of days exposed by the number of days in the period evaluated.
  A PDC≥ 80% is considered as a good adherence to medication.
Percentage of the target cumulative dose of treatment received by the patients | up to 30 months
Influence of factors (yes/no) associated with persistence to AF treatments | up to 30 months
  For a pre-determined list of variables (as defined in the study protocol) in incident AF patients, a multivariate time-dependant Cox model will test several covariates to check if they are associated with persistence to AF treatment.
Number of patients with switch from one AF treatment to the another with no treatment stop | up to 5 years
Number of patients at site of follow-up (identified as 2 lung function tests performed in the center) | up to 5 years
Overall Survival (defined as time from index date (first reimbursement of AF treatment) to death from any cause) | up to5 years
Event-free survival | up to 5 years
  Defined as the time from index date to
  * oxygenotherapy onset
  * hospitalisation for respiratory exacerbations
  * hospitalisation for other respiratory diseases
  * ath from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Clinityx, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com